CLINICAL TRIAL: NCT03284489
Title: Prospective Cohort of Patients With Pancreatitis Hospitalized in West French Intensive Care Units
Brief Title: Post Pancreatitis Complications Study (Based on a Prospective Data Base)
Status: Withdrawn | Type: Observational
Why Stopped: No inclusion
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0207 doublon 2
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Pancreatitis
Keywords: Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients: Patients with pancreatitis
  Interventions: Other: Collection of medical datas from ICU patients

INTERVENTIONS:
Other: Collection of medical datas from ICU patients — Collection of medical datas from ICU patients with pancreatitis on a secured electronic database

SUMMARY:
The purpose of this observational epidemiological study is to investigate the management and the complications associated with pancreatitis. Datas will be analysed to answer pre-defined scientific projects and to improve management of these conditions.

DETAILED DESCRIPTION:
Anonymous datas will be collected by study coordinators in a secured e-database.

Cross audit will be performed to check datas.

ELIGIBILITY:
Inclusion Criteria:

* pancreatitis

Exclusion Criteria:

* consent withdrawal

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pancreatitis hospitalized in ICU
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-04 (Estimated); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
In ICU stay main complications | Within the 28 first days after ICU admission date
  Nosocomial Infections (epidemiology, risk factors, antibiotic susceptibility of pathogens) Organ failures (incidence, risk factors)

SECONDARY OUTCOMES:
Duration of Mechanical Ventilation | During ICU stay (up to 90 days)
Length of ICU stay | During ICU stay (up to 90 days)

OTHER OUTCOMES:
Death | During ICU stay (up to 90 days)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Asehnoune, MD,PhD, Study Chair — Non-Affiliated
Locations (5):
- France (5):
  - Angers University Hospital, Angers
  - Nantes University Hospital, Nantes
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours